CLINICAL TRIAL: NCT07398092
Title: Effects of TRX Suspension Training on Physical Fitness, Gait Performance, and Inflammatory and Growth-Related Biomarkers in Older Men With Sarcopenia: A Randomized Controlled Trial
Brief Title: TRX Suspension Training for Sarcopenia in Older Men
Acronym: TRX-SARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WeiJin Zhang (Other Government)
Responsible Party: Sponsor-Investigator, WeiJin Zhang, Principal Investigator, Sangmyung University
Organization: Sangmyung University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YBU-TRX-SARC-2024-01
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sarcopenia
Keywords: TRX suspension training; Resistance training; Older adults; Physical fitness; Gait performance; Muscle strength; Inflammatory biomarkers; Randomized controlled trial
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to either a TRX suspension training group or a control group and remained in their assigned group throughout the 12-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRX Suspension Training Group (Experimental): Participants assigned to this arm received a supervised TRX suspension training program for 12 weeks. Training sessions were conducted three times per week, with each session lasting approximately 60 minutes. The program included progressive, whole-body resistance exercises targeting the upper limbs, lower limbs, and trunk.
  Interventions: Behavioral: TRX Suspension Training
- Control Group (Other): Participants in the control group maintained their usual daily activities throughout the 12-week study period and did not participate in any structured exercise or training intervention.
  Interventions: Other: Usual Daily Activities

INTERVENTIONS:
Behavioral: TRX Suspension Training — TRX suspension training was delivered as a structured, supervised exercise program conducted three times per week for 12 weeks. Each session lasted approximately 60 minutes and included warm-up, main training, and cool-down phases. The program emphasized progressive, whole-body resistance exercises targeting the upper limbs, lower limbs, and trunk, with training intensity individualized through adjustments in body angle and support points.
  Arms: TRX Suspension Training Group
Other: Usual Daily Activities — Participants continued their usual daily activities during the 12-week study period and did not receive any structured exercise or training intervention.
  Arms: Control Group

SUMMARY:
This randomized controlled trial evaluated the effects of a 12-week TRX suspension training program on physical fitness, gait performance, and selected blood biomarkers in older men with sarcopenia. Sarcopenia is an age-related condition characterized by loss of muscle mass, muscle strength, and physical function, which increases the risk of falls, disability, and reduced quality of life.

A total of 36 older men diagnosed with sarcopenia were randomly assigned to either a TRX suspension training group or a control group. The training group participated in supervised TRX exercise sessions three times per week for 12 weeks, with each session lasting approximately 60 minutes. The control group maintained their usual daily activities without structured exercise intervention.

Physical fitness, walking ability, and blood biomarkers related to inflammation and muscle growth were assessed before and after the intervention. The study aimed to determine whether TRX suspension training is a safe and effective exercise approach for improving muscle strength, balance, walking ability, and biological indicators associated with sarcopenia in older adults.

DETAILED DESCRIPTION:
This study was a single-center, randomized controlled trial designed to examine the effects of TRX suspension training on physical fitness, gait performance, and inflammatory- and growth-related biomarkers in older men with sarcopenia.

Eligible participants were men aged 65 years and older who met established diagnostic criteria for sarcopenia based on low handgrip strength, reduced skeletal muscle mass index, and slow gait speed. After screening, 36 participants were randomly allocated in a 1:1 ratio to either an experimental group receiving TRX suspension training or a control group maintaining usual daily activities.

The intervention consisted of a 12-week TRX suspension training program conducted three times per week. Each training session lasted approximately 60 minutes and included a warm-up period, a main training phase, and a cool-down period. The exercise program emphasized multi-joint, whole-body movements targeting the upper limbs, lower limbs, and trunk. Training intensity and difficulty were progressively adjusted using body angle and support-point principles to ensure safety and individualized progression for older participants.

Assessments were performed before the intervention and within 48 hours after completion of the 12-week program. Outcome measures included physical fitness tests (upper- and lower-limb muscle strength, balance, and agility), gait performance tests (mobility, walking speed, and walking endurance), and fasting blood biomarkers related to inflammation and muscle growth, including interleukin-6, tumor necrosis factor-alpha, insulin-like growth factor-1, C-reactive protein, and vitamin D.

The primary objective of the study was to determine whether TRX suspension training could improve muscle strength and functional mobility in older men with sarcopenia. Secondary objectives included evaluating changes in gait performance and selected biological markers associated with inflammation and muscle metabolism. This study aimed to provide evidence supporting the use of TRX suspension training as a safe and effective exercise strategy for improving physical function and reducing fall risk in older adults with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 65 years or older.
* Diagnosis of sarcopenia based on established criteria, including low handgrip strength, reduced skeletal muscle mass index, and slow gait speed.
* Ability to walk independently without assistive devices.
* Ability to understand the study procedures and provide written informed consent.
* Willingness to participate in the 12-week intervention and complete all required assessments.

Exclusion Criteria:

* Presence of severe cardiovascular disease or other medical conditions that contraindicate moderate-intensity exercise.
* Diagnosis of severe depression, dementia, or other neurological or psychiatric disorders that could interfere with participation.
* Participation in other structured exercise or training programs during the study period.
* History of drug or alcohol abuse.
* Any musculoskeletal, neurological, or systemic condition that would prevent safe participation in the exercise intervention.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Handgrip Strength | Baseline to 12 weeks
  Handgrip strength was measured using a digital handgrip dynamometer. The primary outcome was the change in maximal handgrip strength from baseline to the end of the 12-week intervention period.

SECONDARY OUTCOMES:
Change in 30-Second Chair Stand Test Performance | Baseline to 12 weeks
  Lower-limb muscle strength was assessed using the 30-second chair stand test. The outcome was defined as the change in the number of completed stands from baseline to the end of the 12-week intervention.
Change in 30-Second Arm Curl Test Performance | Baseline to 12 weeks
  Upper-limb muscular endurance was evaluated using the 30-second arm curl test. The outcome was the change in the number of repetitions completed from baseline to the end of the 12-week intervention period.
Change in Single-Leg Stance Time | Baseline to 12 weeks
  Static balance was assessed using the single-leg stance test. The outcome was defined as the change in maximal standing time from baseline to the end of the 12-week intervention.
Change in Four Square Step Test Performance | Baseline to 12 weeks
  Dynamic balance and agility were evaluated using the four square step test. The outcome was the change in completion time from baseline to the end of the 12-week intervention period.
Change in Timed Up and Go Test Performance | Baseline to 12 weeks
  Functional mobility was assessed using the Timed Up and Go test. The outcome was defined as the change in test completion time from baseline to the end of the 12-week intervention.
Change in 10-Meter Walk Test Performance | Baseline to 12 weeks
  Walking speed was evaluated using the 10-meter walk test. The outcome was defined as the change in walking time from baseline to the end of the 12-week intervention period.
Change in Six-Minute Walk Test Distance | Baseline to 12 weeks
  Walking endurance was assessed using the six-minute walk test. The outcome was defined as the change in total walking distance from baseline to the end of the 12-week intervention.
Change in Serum Interleukin-6 Levels | Baseline to 12 weeks
  Systemic inflammation was evaluated by measuring fasting serum interleukin-6 concentrations. The outcome was defined as the change in IL-6 levels from baseline to the end of the 12-week intervention.
Change in Serum Tumor Necrosis Factor-Alpha Levels | Baseline to 12 weeks
  Inflammatory status was assessed by measuring fasting serum tumor necrosis factor-alpha concentrations. The outcome was defined as the change in TNF-alpha levels from baseline to the end of the 12-week intervention.
Change in Serum Insulin-Like Growth Factor-1 Levels | Baseline to 12 weeks
  Muscle anabolic status was assessed by measuring fasting serum insulin-like growth factor-1 concentrations. The outcome was defined as the change in IGF-1 levels from baseline to the end of the 12-week intervention.
Change in Serum Vitamin D Levels | Baseline to 12 weeks
  Vitamin D status was evaluated by measuring fasting serum vitamin D concentrations. The outcome was defined as the change in vitamin D levels from baseline to the end of the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Soo Baek, PhD, Principal Investigator — Department of Sport and Healthcare, Sangmyung University, Seoul, Republic of Korea
Locations (1):
- Yibin University, Yibin, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in the published article, including demographic variables, baseline and post-intervention physical fitness measures, gait performance outcomes, and laboratory biomarker data.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication and will remain available for up to 5 years.
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers who submit a methodologically sound proposal. Requests will be reviewed and approved by the study investigators, and data will be shared upon reasonable request in accordance with applicable ethical and data protection regulations.